CLINICAL TRIAL: NCT03322384
Title: UCDCC#271: A Phase I/II Trial of Epacadostat (Indolamine 2,3 Dioxygenase Inhibitor), Intralesional SD101 (Toll-receptor 9 Agonist), and Radiotherapy in Patients With Advanced Solid Tumors and Lymphoma
Brief Title: UCDCC#271: Phase I/II Trial of Epacadostat, Intralesional SD101, Radiotherapy in Patients With Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Megan Daly, MD, Associate Professor, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1057229; UCDCC#271 (Other: UC Davis IRB)
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumors; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — epacadostat; Radiotherapy

STUDY DESIGN:
Intervention Model Description: All patients will begin epacadostat on day 1 of radiotherapy, which will consist of three threatments over one week. Epacadostat will continue until disease progression or intolerance occurs. On days 1, 8, 15, 22, 29, intralesional injectinons of SD101 will be given to patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): All patients will begin epacadostat on day 1 of radiotherapy, which will consist of three threatments over one week. Epacadostat will continue until disease progression or intolerance occurs. On days 1, 8, 15, 22, 29, intralesional injectinons of SD101 will be given to patients.
  Interventions: Drug: epacadostat; Drug: SD-101; Radiation: Radiotherapy

INTERVENTIONS:
Drug: epacadostat — Epacadostat will be administered orally, in pill form, twice daily until disease progression.
Drug: SD-101 — Four milligrams of SD-101 will be delivered into the treatment lesion by intralesional injection on days 1, 8, 15, 22, and 29.
Radiation: Radiotherapy — Radiotherapy will be delivered to the treatment lesion during the first week of ERS therapy.

SUMMARY:
Checkpoint blockade immunotherapy has revolutionized the management of a variety of advanced malignancies. Monoclonal antibodies targeting the PD-1 / PD-L1 interaction have received FDA approvals for non-small cell lung cancer, melanoma, Merkel cell carcinoma, renal cell carcinoma, hepatocellular, squamous cell carcinoma of the head and neck, microsatellite instability high colorectal carcinoma, urothelial carcinoma, and classical Hodgkin's lymphoma. Despite the promising evidence for deep and durable responses with these agents, the majority of patients either fail to respond or develop resistance to treatment. Thus, there is interested in developing alternative immunotherapeutic strategies. The investigators hypothesize that a novel immunotherapeutic combination of radiotherapy (RT) with intralesional CpG and indolamine-2,3-dioxygenase blockade may offer significant clinical benefit to patients and proposing a microtrial testing this combination for advanced/refractory solid tumors and lymphoma.

DETAILED DESCRIPTION:
Checkpoint blockade immunotherapy has revolutionized the management of a variety of advanced malignancies. Monoclonal antibodies targeting the PD-1 / PD-L1 interaction have received FDA approvals for non-small cell lung cancer, melanoma, Merkel cell carcinoma, renal cell carcinoma, hepatocellular, squamous cell carcinoma of the head and neck, microsatellite instability high colorectal carcinoma, urothelial carcinoma, and classical Hodgkin's lymphoma. Despite the promising evidence for deep and durable responses with these agents, the majority of patients either fail to respond or develop resistance to treatment. Thus, there is interested in developing alternative immunotherapeutic strategies. The investigators hypothesize that a novel immunotherapeutic combination of radiotherapy (RT)with intralesional CpG and indolamine-2,3-dioxygenase (IDO) blockade may offer significant clinical benefit to patients and proposing a microtrial testing this combination for advanced/refractory solid tumors and lymphoma.

Unmethylated CpG DNA is a component bacterial genomes and is the agonist of Toll Like Receptor-9, an endosomal pattern recognition receptor of antigen presenting cells. TLR9 activation results in downstream production of IFN-α, interleukin-6 interleukin-12. These cytokines induce naive T cells to differentiate to helper T cells. CpG has demonstrated significant synergy with radiotherapy to induce regression of refractory systemic and cutaneous lymphomas both within radiation treatment field and un-irradiated metastases. SD-101 is a synthetic oligodeoxynucleotide enriched with CpG motifs.

IDO is an enzyme that converts the essential amino acid tryptophan to kynurenine. The availability of tryptophan is essential to sustaining both helper T cell and effector T cell activation. Overexpression of IDO by tumor cells or antigen presenting cells serves to arrest T cell activation thus acting as an immunosuppressive enzyme. Epacadostat (INCB024360) is an inhibitor of the enzyme indoleamine 2,3-dioxygenase 1 (IDO1) that has shown promise in the treatment of solid tumors and lymphomas in ongoing Phase I/II studies.

The investigators have shown in animal studies that IDO upregulation limits tumor response to RT + CpG and that addition of IDO blockade improves therapeutic efficacy. On the basis of these data, the investigators hypothesize that IDO inhibition will improve upon the known historical efficacy of RT + CpG therapy, and will be highly effective and well tolerated in the management of advanced solid tumors and lymphomas.

This is a phase I/II study. For the phase I portion the primary endpoint is to determine the maximum tolerated dose of epacadostat in combination with radiotherapy and SD-101. For the phase II portion the primary endpoint is safety and toxicity per CTCAE v4.03 criteriae. The secondary endpoint is the abscopal response rate defined as the objective response rate at un-irradiated lesions per irRECIST criteria.

Up to three dose levels of epacadostat will be evaluated: 100 mg bid, 200 mg bid and 300 mg bid each day of the study. Radiotherapy will be delivered to the treatment lesion during the first week using standard-of-care palliative fractionation regimens of 8 Gy x 3 fractions, 4 Gy x 5 fractions, or 2 Gy x 2 fractions. Four milligrams of SD-101 will be delivered into the treatment lesion by intralesional injection on days 1, 8, 15, with optional additional injections on days 22, and 29. On Day 1, biopsy will precede intralesional injection, RT, or epacadostat. Intralesional injections will be performed by palpation of the lesion or under ultrasound or CT guidance as indicated. CT response assessments and labs will be performed every 60 days. Patients will continue on epacadostat until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >18 years of age with histologically proven solid malignancy, high-grade lymphoma or low-grade lymphoma.
2. Patients with incurable, advanced or metastatic disease refractory to at least one previous line of standard of care therapy.
3. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 - 2 (Appendix 1).
4. Presence of a candidate treatment lesion (subcutaneous, nodal, or visceral) accessible and safe for radiotherapy and serial intralesional injections as specified by the protocol.
5. Presence of at least one target lesion (distinct from treatment lesion and outside of treatment lesion radiation field) evaluable for response by irRECIST.
6. 14 day wash-out period from any previous chemotherapy, targeted therapy or radiotherapy, 21 day washout period from previous immunotherapy.
7. Life expectancy ≥ 6 months.
8. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days of the first study treatment:

   o ANC > 1500 cells/ul; WBC count > 2500/uL; Lymphocyte count >500/uL; Platelet count > 100,000/uL; Hemoglobin > 9 g/dL
9. Liver function tests meeting one of the following criteria:

   1. AST and ALT < 2.5 x ULN with alkaline phosphatase < 2.5 x ULN OR
   2. AST and ALT < 1.5 x ULN, with alkaline phosphatase > 2.5 x ULN
   3. Serum bilirubin < 1.0 x ULN. Direct bili < 40% if total bili > ULN in patients with Gilbert's syndrome.
10. INR and aPTT < 1.5 x ULN.
11. Serum Cr < 1.5 X ULN or CrCl > 50 ml/min.
12. No active auto-immune disease and not on therapy for auto-immune disease. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible. Patients who have adrenal insufficiency and hypophysitis from prior immunotherapy if they are on stable medical replacement doses are eligible.
13. No other active malignancy.
14. Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible.
15. For female patients of childbearing potential and male patients with partners of childbearing potential agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for 6 months after trial completion.
16. Signed informed consent.
17. At least 9 months from stem cell transplant with no active graft versus host disease.
18. Ability to comply with the protocol.

Exclusion Criteria:

1. Uncontrolled concomitant disease that in the opinion of the investigator would interfere with the patient's safety or compliance on trial.
2. Significant cardiovascular disease (NYHA Class II or greater); myocardial infarction within 3 month prior to randomization, unstable arrhythmias, unstable angina or a patient with a known LVEF (Left Ventricular Ejection Fraction) < 40%
3. Severe infection that in the opinion of the investigator would interfere with the patients safety or compliance on trial within 2 weeks prior to enrollment. Oral or IV antibiotics within 2 weeks or 5 half-lives prior to enrollment.
4. Active tuberculosis
5. History of severe autoimmune disease that in the opinion of the investigator would interfere with patient safety or compliance on trial.
6. Positive for Human Immunodeficiency Virus (HIV), Hepatitis B (Hepatitis B Surface Antigen [HBsAg] reactive), or Hepatitis C virus (Hepatitis C Virus Ribonucleic Acid [HCV RNA] (qualitative) is detected)
7. Previous treatment with epacadostat, SD-101, or any other IDO inhibitor or CpG molecule.
8. Treatment with systemic corticosteroids or other systemic immunosuppressive medications within past 4 weeks or 5 half-lives whichever is shorter. Use of inhaled or topical steroids or systemic corticosteroids < 10 mg/ day of prednisone (or equivalent) is permitted.
9. Pregnant and/or lactating women.
10. Evidence of active interstitial lung disease or active non-infectious pneumonitis
11. Receipt of live attenuated vaccine within 30 days before the first dose of study treatment.
12. Use of any UGT1A9 inhibitor while on active study treatment, including the following: diclofenac, imipramine, ketoconazole, mefenamic acid, and probenecid.
13. Known allergy or reaction to any component of either study drug formulation.
14. Subjects receiving Monoamine Oxidase Inhibitors (MAOIs) or drug which has significant MAOI activity (meperidine, linezolid, methylene blue) from 21 days prior to Day 1 through 2 weeks after the final dose of epacadostat has been administered.
15. Any history of Serotonin Syndrome (SS) after receiving serotonergic drugs.
16. Known contraindications to radiotherapy including but not limited to radiation sensitivity syndromes such as xeroderma pigmentosum and ataxia telangiectasia mutated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Daly, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 20
Completed | 14
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: To determine the maximum tolerated dose (MTD) of epacadostat that can be given with radiotherapy and intralesional SD-101 immunotherapy for the phase I portion of the study. The MTD will be determined using a standard 3+3 design. Patients will be monitored weekly during a 30-day dose-limiting toxicity (DLT) period. MTD can be defined as The maximum dose at which <2 of 6 patients experienced a DLT.
Time Frame: Up to 30 days of treatment
Measure: Number; unit: mg
Arm/Group | Experimental
Number analyzed (Participants) | 6
mg | 300

2. Primary Outcome: Incidence of Related Adverse Events [Safety and Tolerability]
Description: To characterize the safety profile of this regimen using CTCAE v4.03 (Common Toxicity Criteria for Adverse Events version 4.03) in the phase II expansion . The expansion phase (phase II) will be conducted using the MTD defined as the highest dose at which no more than one of six patients develops a DLT or Dose Level 1 if the MTD is not reached. Patients will be monitored every week during the first 30 days of study and then monthly thereafter up to a period of 1 year.
Time Frame: Through study completion, an average of one year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 20
Participants | 17

3. Secondary Outcome: Abscopal Response Rate
Description: Abscopal Response Rate (ARR) is defined as objective response rate (the percentage of patient that achieve a partial or complete response) at unirradiated sites using irRECIST criteria using imaging obtained every 60 days during the 1 year study period.
Time Frame: Through study completion, an average of one year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 14
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 1 year.
Description: Incidence of Treatment-Emergent Adverse Events according CTCAE v4.03
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 10/20
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=20)
Gastrointestinal disorders - Other, specify: lower GI bleed (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Investigations - Other, specify: transanimitis (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify: electrolyte and fluid disorder (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify:disease progres (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=20)
Anemia (Blood and lymphatic system disorders) | 5
Sinus tachycardia (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 9
Chills (General disorders) | 2
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 11
Injection site reaction (General disorders) | 5
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 4
Creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 7
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Paresthesia (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03322384/Prot_SAP_000.pdf